CLINICAL TRIAL: NCT02407353
Title: A Phase 1 Investigator-and-subject Blind, Randomized, Placebo Controlled, Parallel Study In Healthy Subjects To Evaluate The Pharmacodynamic Effects Of Single Oral Doses Of Pf-06648671 On Aβ Concentrations In Cerebrospinal Fluid Using Serial Sampling Methodology
Brief Title: A Study to Evaluate the Pharmacodynamic Effects of Single Oral Doses of PF-06648671 on β-Amyloid (Aβ) Concentrations in Cerebrospinal Fluid (CSF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7991003
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Subjects
Keywords: Phase 1; Double blind; Placebo-Controlled; Parallel Design; CSF Aβ Concentrations; PF-06648671

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-06648671 High dose group (Experimental): subjects receive a single oral dose of PF-06648671 at 300 mg
  Interventions: Drug: PF-06648671
- PF-06648671 Low dose group (Experimental): Subjects receive a single oral dose of PF-06648671 lower than 300 mg dose
  Interventions: Drug: PF-06648671
- Placebo group (Placebo Comparator): Subjects receive matching placebo
  Interventions: Drug: Placebo
- PF-06648671 Low dose group (2) (Experimental): Optional arm. Subjects receive a single oral dose of PF-06648671 at second lower dose if 300 mg dose is not repeated in cohort 2
  Interventions: Drug: PF-06648671

INTERVENTIONS:
Drug: PF-06648671 — Experimental Pfizer compound which will be dosed as oral suspension, single dose at 300 mg and/or 1-2 lower doses
  Arms: PF-06648671 High dose group; PF-06648671 Low dose group; PF-06648671 Low dose group (2)
Drug: Placebo — Placebo which will be dosed as oral suspension, single doses to match PF-06648671
  Arms: Placebo group

SUMMARY:
This is phase 1 investigator-and-subject blind, sponsor open, randomized, placebo controlled, parallel study in healthy subjects to evaluate the pharmacodynamics effect of single oral doses of PF-06648671 on CSF Aβ concentrations using serial CSF sampling methodology.

DETAILED DESCRIPTION:
This study is investigator-and-subject blind, sponsor open, randomized, placebo-controlled, parallel study in healthy subjects to evaluate central (CSF) and peripheral (plasma) pharmacodynamics effects (Abeta) over 36 hours post single doses of PF-06648671. Two cohorts will be run in sequential. the first cohort is to evaluate the Abeta effect at top dose of 300 mg PF-06648671 and second cohort is to evaluate the Abeta effect at top dose (if more subjects are required) and/or 1-2 lower doses

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential
* BMI of 17.5 to 30.5 kg/m2 and a total body weight >50 kg (110 lbs)
* Evidence of a personally signed and dated informed consent document indicating that subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated asymptomatic, seasonal allergies at the time of dosing)
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication (whichever is longer)
* Subjects with a history of significant active bleeding, coagulation disorder or clinically significant finding on prothrombin time/ partial thromboplastin time/International Normalized Ratio (PT/PTT/INR) at Screening
* Subjects with lower spinal malformations (on physical examination), local spinal infection, or other abnormalities that would exclude puncture (LP)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
CSF Aβ40 and Aβ42 concentration at maximum change from baseline | 0-36 hours postdose

SECONDARY OUTCOMES:
Number of participants with AEs and SAEs | 0-2 weeks
  Counts of participants who have TEAEs, defined as newly occuring or worsening after first dose. Relatedness to PF-06648671 will be assessed by the investigator (Yes/No). Participants with multiple occurrence of an AE within a category will be counted once within the category
supine vital sign | 0-2 weeks
  Measurement of supine vital signs
Electrocardiogram (ECG) | 0-2 weeks
  Measurement of standard 12-lead ECG (single)
Maximum Observed Plasma Concentration (Cmax) | 0-72 hours postdose
Area Under the Curve from Time Zero to Last Quantifiable Plasma Concentration (AUClast) | 0-72 hours postdose
Area Under the Curve From Time Zero to Extrapolated Infinite Time in Plasma (AUCinf) | 0-72 hours postdose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-72 hours postdose
Plasma Decay Half-life (t1/2) | 0-72 hours postdose
Apparent Oral Clearance (CL/F) | 0-72 hours postdose
Apparent Volume of Distribution (Vz/F)) | 0-72 hours postdose
Maximum Observed CSF Concentration (CSF Cmax) | 0-36 hours postdose
Area Under the Curve from Time Zero to Last Quantifiable Concentration in CSF (CSF AUClast) | 0-36 hours postdose
Area Under the Curve From Time Zero to Extrapolated Infinite Time in CSF (CSF AUCinf) | 0-36 hours postdose
CSF Decay Half-life (CSF t1/2) | 0-36 hours postdose
Plasma Aβ40, Aβ42 and Aβtotal | 0-72 hours postdose
  Plasma Aβ40, Aβ42 and Aβtotal if possible
CSF Aβ37, Aβ38 and Aβtotal Concentration | 0-36 hours postdose
Number of participants with lab test values of potential clinical importance | 0-2 weeks
  Pre-defined criteria were established for each lab test to identify potential clinical importance

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - California Clinical Trials Medical Group, Inc., Glendale, California
  - Glendale Adventist Medical Center, Glendale, California

REFERENCES:
- [Derived] Ahn JE, Carrieri C, Dela Cruz F, Fullerton T, Hajos-Korcsok E, He P, Kantaridis C, Leurent C, Liu R, Mancuso J, Mendes da Costa L, Qiu R. Pharmacokinetic and Pharmacodynamic Effects of a gamma-Secretase Modulator, PF-06648671, on CSF Amyloid-beta Peptides in Randomized Phase I Studies. Clin Pharmacol Ther. 2020 Jan;107(1):211-220. doi: 10.1002/cpt.1570. Epub 2019 Sep 11. PMID 31314925
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7991003&StudyName=A%20Phase%201%20Investigator-and-subject%20Blind%2C%20Randomized%2C%20Placebo%20Controlled%2C%20Parallel%20Study%20In%20Healthy%20Subjects%20To%20Evaluate%20The%20Pharmacodynamic%20Effects%20Of%20Single%20Oral%20Doses%20Of%20Pf-06648671%20On%20A%CE%B2%20Concentrations%20In%20Cerebrospinal%20Fluid%20Using%20Serial%20Sampling%20Methodology